CLINICAL TRIAL: NCT07382817
Title: A Phase 1 Safety and Efficacy Study of JV-394 Autologous Anti-CD94 Chimeric Antigen Receptor T Cell Therapy in Patients With Relapsed or Refractory CD94+ T/NK Cell Neoplasms
Brief Title: Phase 1 Study of JV-394 Autologous Anti-CD94 CAR T for r/r CD94+ T/NK Cell Neoplasms
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1446; NCI-2026-00809 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2026-01-30; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms
Keywords: CAR T cell therapy; T Cell Lymphoma; T/NK-Cell Lymphoma
MeSH Terms: conditions — Neoplasms; Lymphoma, T-Cell; Lymphoma, Extranodal NK-T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment with JV-394 CAR T (Experimental): Infusion of JV-394 and subsequent safety monitoring will be conducted at a healthcare facility. Participants may be hospitalized for JV-394 infusion and subsequent safety monitoring at the discretion of the investigator or treating physician. JV-394 will be administered as a single infusion of anti-CD94 CAR-transduced autologous T cells on day 0 in under 30 minutes.
  Interventions: Drug: JV-394

INTERVENTIONS:
Drug: JV-394 — Given by infusion

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of JV-394 (a type of autologous CAR-T cell therapy) that can be given to patients who have T/NK cell lymphoma that is relapsed or refractory. The safety and possible side effects of JV-394 will also be studied.

DETAILED DESCRIPTION:
Primary Objective:

The primary objective is to determine the safety and identify the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of JV-394 in patients with CD94+ r/r T/NK cell malignancies.

Secondary Objective:

The secondary objectives are to determine the efficacy in adults with r/r CD94+ T/NK cell malignancies at the MTD or RP2D of JV-394. Secondary end points include overall response rate (ORR; including CR+PR) and CR rate as defined by Lugano or Olsen Criteria, duration of response (DOR), progression free survival (PFS) and overall survival (OS).41,42

Exploratory Objective:

The exploratory objectives are to assess the cellular kinetics and pharmacodynamic effects of JV-394 anti-CD94 CAR T cell product and to evaluate biomarkers associated with response, resistance, and toxicity after administration of CAR T product in blood and tumor samples.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age.
2. Confirmed T/NK cell malignancies as per local histopathological assessment.
3. Relapsed or refractory disease after at least one line of systemic therapy or intolerant to standard therapy for their cancer.
4. Eligible histologies include: extranodal NK/TCL, hepatosplenic TCL, primary cutaneous CD8+ aggressive epidermotropic cytotoxic TCL, subcutaneous panniculitis-like TCL, monomorphic epitheliotropic intestinal TCL, enteropathy-associated TCL, primary cutaneous γδ TCL, peripheral TCL cytotoxic type, Epstein-Barr virus (EBV)+ nodal T/NK cell lymphoma, and other CD94+ T/NK cell malignancies not listed above.
5. ≥50% of tumor cells are positive for CD94 by flow cytometry or IHC. Historical documentation of CD94 expression in the tumor is acceptable if available. If there is no historical documentation of CD94 expression, testing of archival tumor tissue or fresh tumor biopsy is required. Testing of archival tumor tissue may be done by IHC following a prescreening consent.
6. At least two weeks or 5 half-lives, whichever is shorter, must have elapsed since any prior systemic anti-cancer therapy or 1 week from prior radiation therapy prior to leukapheresis.
7. ECOG performance status of 0-1 (Appendix 1).
8. For non-cutaneous lymphomas, at least one measurable lesion as per Lugano 2014 classification. Subjects with primary cutaneous variants must have at least 1 measurable lesion that is evaluable using the Olsen 2021 criteria.
9. Toxicities due to prior therapy must be stable and recovered to ≤grade 1 (except for clinically non-significant toxicities such as alopecia).
10. Absolute neutrophil count of ≥1.0×109 /L.
11. Absolute lymphocyte count of ≥0.1×109 /L.
12. Platelet count of ≥75×109 /L.
13. Creatinine clearance (as estimated by Cockcroft Gault) ≥45 mL/min.
14. Serum alanine transaminase (ALT) / aspartate transaminase (AST) ≤5 times the upper limit of normal (ULN).
15. Total bilirubin ≤2 mg/dL, except in patients with Gilbert's syndrome.
16. Cardiac ejection fraction ≥45% with no evidence of clinically significant pericardial effusion.
17. Baseline oxygen saturation ≥92% on room air.
18. Women of childbearing potential must have a negative serum or urine pregnancy test (women who have had hysterectomy and women who are over the age of 45 years and have not had a menstrual period for at least 1 year are not considered to be of childbearing potential).

Exclusion Criteria:

1. Subjects with aggressive NK cell leukemia and indolent T/NK cell malignancies such as TLGL or NK-LGL.
2. Patients with tumor cells in the peripheral blood ≥1% of lymphocytes as determined by flow cytometry.
3. Active central nervous system (CNS) lymphoma including patients with detectable cerebrospinal fluid malignant cells or brain metastases. Patients with prior CNS lymphoma that has been effectively treated will be eligible if treatment was completed at least one year prior to enrolment and there is no evidence of disease on MRI with gadolinium contrast at the time of screening.
4. Autologous stem cell transplantation within 6 weeks.
5. Allogeneic cell transplantation within 3 months or active graft versus host disease.
6. History of any form of primary immunodeficiency that in the opinion of the investigator may affect efficacy of the CAR T product.
7. History of any one of the following cardiovascular conditions within the past 6 months: Class III or IV heart failure as defined by the New York Heart Association, cardiac angioplasty or stenting, myocardial infarction, unstable angina, or other clinically significant cardiac disease.
8. History of malignancy other than nonmelanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast) unless disease free for at least 2 years and treated with curative intent. Patients with a prior history of malignancy whose natural history or treatment (e.g. hormonal therapy) does not have the potential to interfere with either the safety or efficacy assessment of the investigational regimen in the opinion of the investigator may be included.
9. Presence of fungal, bacterial, viral, or other infection that is uncontrolled or requiring intravenous antimicrobials for management. Simple urinary tract infection and uncomplicated bacterial pharyngitis or localized skin infections are permitted if responding to active treatment and after consultation with the Principal Investigator.
10. Known history of infection with HIV or hepatitis B (HBsAg positive) or hepatitis C virus (anti-HCV positive). A history of hepatitis B or hepatitis C is permitted if the viral load is undetectable per quantitative PCR and/or nucleic acid testing.
11. Active autoimmune (e.g. Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus) or inflammatory disease (including graft-versus-host disease) requiring systemic immunosuppressive therapy. Physiological replacement of corticosteroids of up to 7.5 mg of prednisone or equivalent per day, and topical and inhaled corticosteroids are permitted.
12. History or presence of CNS disorders such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement.
13. Patients with cardiac atrial or cardiac ventricular lymphoma involvement.
14. Requirement for urgent therapy due to tumor mass effect such as bowel obstruction or blood vessel compression.
15. Any medical condition likely to interfere with assessment of safety or efficacy of study treatment.
16. Live vaccine ≤6 weeks prior to planned start of conditioning regimen.
17. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the conditioning chemotherapy on the fetus or infant.
18. Females of childbearing potential and males of child fathering potential who are not willing to practice two methods of birth control from the time of consent through 6 months after infusion of the study drug.
19. In the investigator's judgment, the patient is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation.
20. Patients who are receiving any other investigational agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2029-12-09 (Estimated); Study Completion 2031-12-09 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Sattva S Neelapu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org